CLINICAL TRIAL: NCT06454175
Title: A Randomised, Double-blind, Placebo-controlled Phase I Clinical Trial to Evaluate the Safety and Tolerability of 15-valent Human Papillomavirus Recombinant Vaccine (Hansenulapolymorpha) in Healthy Chinese People Aged 18-45 Years
Brief Title: A Phase I Clinical Trial to Evaluate the Safety of 15-valent HPV Vaccine in Healthy Chinese People Aged 18-45 Years
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Bovax Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 15-HPV-1001
Record Dates: First submitted 2024-06-06; First posted 2024-06-12 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-06

CONDITIONS: HPV Infection; HPV-Related Carcinoma; Genital Wart; HPV-Related Intraepithelial Neoplasia
MeSH Terms: conditions — Papillomavirus Infections; Condylomata Acuminata

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HPV-vaccine group (Experimental): According to the 0, 2, and 6 months immunization schedule, intramuscular injection of the upper arm deltoid muscle, 3 doses of the 15-HPV vaccine
  Interventions: Biological: 15-valent recombinant human papillomavirus vaccine (Hansenulapolymorpha)
- Placebo group (Placebo Comparator): According to the 0, 2, and 6 months immunization schedule, intramuscular injection of the upper arm deltoid muscle, 3 doses of the placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Placebo — immunization schedule：Month 0，Month 2，Month 6
  Arms: Placebo group
Biological: 15-valent recombinant human papillomavirus vaccine (Hansenulapolymorpha) — immunization schedule：Month 0，Month 2，Month 6
  Arms: HPV-vaccine group

SUMMARY:
To evaluate the safety and tolerability of 15-valent HPV vaccine in 9-45year-old participants.

DETAILED DESCRIPTION:
A phase 1 random, double blind, placebo control trail was plan to conducted in 72 healthy participants in the 2 age groups(18-45 years old and 9-17 years old). The 72 subjects to be inoculated with middle and high dose vaccine first in sequence if there was no safety issue.

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged 9-45；
2. Participans aged 18-45 who can provide legal identification，participants aged 9-17 and their guardian can provide legal identification；
3. Participants and/or their guardian sign an informed consent form (a 9-17 year old participant signs an informed notification);
4. Axillary temperature was less than 37.3 ℃（>14 years old）or less than 37.5℃（≤14 years old）at the time of enrollment；
5. Be able to comply with study protocol requirements；
6. Women were not pregnant at the time of enrollment (negative blood pregnancy test), did not have lactation period，had no birth plan within the 30 days after receiving the whole vaccination;
7. Women with reproductive age take effective contraceptive measures within 2 weeks before enrollment in the study;
8. Agree to take effective contraceptive measures within 30 days after receiving the whole vaccination (effective contraceptives include: oral contraceptives, injection or embedding contraceptives, sustained release topical contraceptives, hormone patches, intrauterine devices), sterilization, abstinence, condoms (male), diaphragms, cervical caps, etc.
9. Women who receiving hormone test has a regular menstruation for more than one year

Exclusion Criteria:

1. Have been vaccinated with other HPV vaccines or planned to vaccinate other HPV vaccines during the study period；
2. Plan to participate other clinical trials during the study period，or participated other clinical trials within 3 months before enrollment, including vaccine or drug;
3. Before the first dose is vaccinated, the laboratory test indicators specified in the program are abnormal, except for NCS determined by the clinician;
4. History of CIN2/AIS/Cervical Cancer/Pelvic radiation therapy;
5. History of HPV-related external genital diseases (such as genital warts, Vulvar intraepithelial neoplasia, Vaginal intraepithelial neoplasia, Penis/perianal/perineum intraepithelial neoplasia, Penile/perianal/perineal cancer) 、anal intraepithelial neoplasia and related cancer, or head and neck cancer；history of sexually transmitted diseases (including syphilis， Gonorrhea, genital chlamydia infection, genital herpes, soft chancre, sexually transmitted lymphogranuloma, inguinal granuloma, etc.);
6. Has been diagnosed as having congenital or acquired immunodeficiency, human immunodeficiency virus (HIV) infection, lymphoma, leukemia, systemic lupus erythematosu, rheumatoid arthritis, juvenile Rheumatoid arthritis, Pernicious Anemia, Ulcerative colitis or other autoimmune conditions (such as Type 1 diabetes, Graves' disease, hashimoto thyroiditi, etc.);
7. History of convulsions, epilepsy, except of febrile convulsions in children 5 years of age and younger;
8. History of severe allergy that requires medical intervention, including but not limited to severe adverse reactions caused by vaccine or drug, eg anaphylactic shock, allergic laryngeal edema, allergic purpura, thrombocytopenia sexual purpura, local allergic necrosis (Arthus reaction), widespread urticaria, dyspnea, angioedema, etc.; History of severe side effect caused by vaccination or severe allergy to any of the components of the investigational vaccine, including histidine, sodium chloride, aluminium phosphate, Polysorbate 80 and water for injection;
9. Suffering from severe cardiovascular disease, severe liver and kidney disease, malignant tumor, and serious infectious disease, such as: tuberculosis, viral hepatitis, etc.;
10. Before the enrollment, the physical examination was untreatment or uncontrolled hypertension, (18-45 year olds: systolic blood pressure ≥140mmHg and / or diastolic blood pressure ≥90mmHg, 9-17 year olds: systolic blood pressure ≥120mmHg and / or diastolic blood pressure ≥80mmHg);
11. Coagulation disorders: such as Congenital or acquired hemophilia, Coagulation factor deficiency, clotting disorders, thrombocytopenia, etc.;
12. No spleen or functional spleen, and no spleen caused by any condition;
13. Receive any Immunosuppressive therapy product within 1 month prior to the first vaccination, or plan to receive such product from Day 0 to Month 7 (30 days after receiving the third dose of vaccination)，e.g. systemic medication for glucocorticoid (>20mg/day or 2mg/kg/day, continuous use ≥2 weeks), but local medication can be used (such as ointment, eye drops, inhalants) Or nasal spray);
14. Receive any immunoglobulin or blood product within 3 months prior to the first injection, or plan to receive such product from Day 0 to Month 7 (30 days after receiving the third dose of vaccination);
15. 3 days before vaccination, suffering from acute illness or acute exacerbation of chronic disease; using fever reducer, Antihistamines, and Analgesics(such as: Acetaminophen, Ibuprofen, Aspirin, loratadine, Cetirizine, etc. )
16. Receiving inactivated vaccine or recombinant vaccine or live-attenuated vaccine or nucleic acid vaccine or adenovirus vaccine within 14 days before vaccination;
17. History of mental disorders or family history of mental health disorder (immediate family)
18. Plan to move out of the city before the end of the study or leave the local area for a long time during the scheduled study visit;
19. The investigator believes that the participant has any condition that may interfere with the assessment of the purpose of the study.

Ages: 9 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-08-03 (Actual); Primary Completion 2025-02-05 (Estimated); Study Completion 2025-07-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Adverse Events | Up to 30 minutes after any vaccination
  AE of local and systemic reactions within 30 minutes after each dose
Percentage of Participants With Solicited Adverse Events | Up to 14 days after any vaccination
  The percentage of participants with one or more solicited AEs was assessed.
Percentage of Participants With Unsolicited Adverse Events | Up to 30 days after any vaccination
  The percentage of participants with one or more unsolicited AEs was assessed.
Percentage of Participants With Serious Adverse Events | From Day 0 after the first dose of vaccination to 6 months after the thrid dose
  The percentage of participants with one or more SAEs was assessed
Percentage of Female Participants With Pregnancy Events | From Day 0 after the first dose of vaccination to 6 months after the thrid dose
  The percentage of participants with Pregnancy Events was assessed

CONTACTS AND LOCATIONS:
Overall Officials: LIRONG HUANG, Master, Principal Investigator — Guangxi Center for Disease Prevention and Crontrol
Locations (1):
- Guangxi Zhuang Autonomous Region Center for Disease Control and Prevention, Guangxi, China

IPD SHARING:
Plan to Share IPD: No